CLINICAL TRIAL: NCT00908713
Title: Corticoids in Severe Community-acquired Pneumonia
Brief Title: Corticoids in Severe Community-Acquired Pneumonia (CAP)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Carlos Agusti, Consultor Senior, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FIS 2003-CA
Record Dates: First submitted 2009-05-26; First posted 2009-05-27 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2013-03

CONDITIONS: Community-Acquired Pneumonia
Keywords: Severe CAP; Adjuvant therapy; Glucocorticoids; CAP Fine V with C-reactive protein >= 15 mg/100 mL
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Methylprednisolone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- methylprednisolone (Experimental): methylprednisolone 0.5 mg/kg body weight every 12 h for 5 days
  Interventions: Drug: methylprednisolone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: methylprednisolone — methylprednisolone 0.5 mg/kg body weight every 12 h for 5 days
  Other Names: solumoderin
  Arms: methylprednisolone
Drug: Placebo — Sodium chloride 0.9% 10 mL every 12 h for 5 days
  Other Names: sodium chloride
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy of glucocorticoids as an adjuvant therapy in patients with severe community-acquired pneumonia (CAP) (Fine V). The hypothesis of the study is that glucocorticoids can modulate the excessive inflammatory response in patients with severe CAP without any significant side effects, showing a benefit in the percentage of non-response to the empiric antimicrobial treatment.

DETAILED DESCRIPTION:
Community acquired pneumonia (CAP) is associated with a local and systemic inflammatory response conducted by different pro and counter inflammatory cytokines. The evolution of the infection is mainly dependent on the intensity of the inflammatory response. The AIM of the project is to determine the clinical usefulness of methylprednisolone treatment (0,5 mg/ Kg weight every 12h for 5 days in patients with severe CAP and an excessive inflammatory response( patients identified based on a cut-off point of the reactive C protein (RCP) of 15 mg/dl). A randomized double blind placebo controlled study with two arms will be performed: The study group (patients with excessive inflammatory response) will receive methylprednisolone + antibiotics. Control group will receive placebo + antibiotics. Patients older than 18 years with Fine V pneumonia will be recruited. Clinical data and prognostic factors (APACHE II and, SOFA scores, etiology, mortality at ICU and at 28 days) will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Severe community-acquired pneumonia Fine V
* CRP >=15 mg/100 mL

Exclusion Criteria:

* Major contraindications for corticosteroids, such as uncontrolled diabetes, immunosuppression
* Previous glucocorticoid treatment during the previous month
* Documented extrapulmonary infection
* Previous hospitalization in the previous month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2004-01; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Rate of non-response to empiric antimicrobial treatment | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Agusti, MD, Principal Investigator — Hospital Clinic, Barcelona,Spain.
Locations (3):
- Spain (3):
  - Servei Pneumologia. Hospital Clinic, Barcelona, Catalonia
  - Servei Pneumoloiga. Hospital Clinic, Barcelona, Catalonia
  - Hospital Clinic, Barcelona

REFERENCES:
- [Derived] Ceccato A, Cilloniz C, Ranzani OT, Menendez R, Agusti C, Gabarrus A, Ferrer M, Sibila O, Niederman MS, Torres A. Treatment with macrolides and glucocorticosteroids in severe community-acquired pneumonia: A post-hoc exploratory analysis of a randomized controlled trial. PLoS One. 2017 Jun 15;12(6):e0178022. doi: 10.1371/journal.pone.0178022. eCollection 2017. PMID 28617807
- [Derived] Torres A, Sibila O, Ferrer M, Polverino E, Menendez R, Mensa J, Gabarrus A, Sellares J, Restrepo MI, Anzueto A, Niederman MS, Agusti C. Effect of corticosteroids on treatment failure among hospitalized patients with severe community-acquired pneumonia and high inflammatory response: a randomized clinical trial. JAMA. 2015 Feb 17;313(7):677-86. doi: 10.1001/jama.2015.88. PMID 25688779
- See also: Related Info — http://www.idibapsrespiratoryresearch.org/